CLINICAL TRIAL: NCT03651310
Title: The Effect of Music Listening on Preoperative Anxiety in Female Pelvic Medicine and Reconstructive Surgery: A Randomized Trial
Brief Title: Music Listening on Preoperative Anxiety in Female Pelvic Medicine and Reconstructive Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Thythy Pham, MD, Assistant Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 211003
Record Dates: First submitted 2018-08-23; First posted 2018-08-29 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Preoperative Anxiety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): waiting in preoperative area without music listening.
- Music Listening Group (Active Comparator): The music listening group will be given a set of noise canceling headphones and an MP3 player with multiple tracks representing different music genres to use while in preoperative area.
  Interventions: Other: Music Listening Group

INTERVENTIONS:
Other: Music Listening Group — Waiting in preoperative area with music listening.
  Arms: Music Listening Group

SUMMARY:
Can music listening decrease a patient's anxiety before surgery? The investigators hypothesize that music listening will decrease a patient's pre-operative anxiety significantly more than no music listening.

The investigators aim to see if additional variables affect a patient's anxiety and response to music listening, such as demographic factors (age, race, prior surgical experience, type of surgery planned) and music background (experience playing a musical instrument, music listening habits). The investigators also aim to see if pre-operative music listening is associated with improved patient satisfaction.

DETAILED DESCRIPTION:
Does music listening decrease preoperative anxiety in women who are scheduled for pelvic reconstructive surgery? Participants will be approached on the day of pelvic reconstructive surgery while they wait in the pre-operative area for surgery. For the sake of not disrupting the flow of the surgery schedule, patients will be consented approximately 45 minutes before the anticipated start time of surgery. If patient agrees to participate, they will be consented and evaluated for eligibility. Once informed consent is obtained, the patient will be randomized to either the music listening group or the control group. All patients will be asked to complete a STAI-Y1 and demographics questionnaire while awaiting surgery. Those in the music listening group will be asked to answer additional questions regarding their background and experience with music.

Control group:

Participants in the control group will complete another STAI-Y1 questionnaire after 30 minutes of waiting. At the patient's routine 6 weeks postoperative visit, she will be asked to rate her overall satisfaction with her surgery and her satisfaction with the preoperative experience.

Music listening group:

The music listening group will be given a set of noise canceling headphones and an MP3 player with multiple tracks representing different music genres to use while in preoperative area. Patients will be given a handout listing the music genre types and asked to circle which music type they listened to during the study. Genre types include classical instrumental, classical piano, smooth jazz, gospel, and new age. After 30 minutes, patients will be asked to complete another STAI-Y1 questionnaire. They will be given the option to continue listening to music up until the time of surgery; however no additional STAI-Y1 questionnaires will be administered. Headphones and the MP3 player will be taken from the patient as she is being transported to the operating room. The headphones and MP3 player will be cleaned with alcohol wipes and reused for other participants in the study.

At the patient's routine 6 weeks postoperative visit, she will be asked to rate her overall satisfaction with her surgery, her satisfaction with the preoperative experience, and whether she would recommend pre-operative music listening to others.

ELIGIBILITY:
Inclusion Criteria:

* Women who are patients of the Loyola University Medical Center Division of Female Pelvic Medicine and Reconstructive Surgery and are scheduled for pelvic reconstructive surgery.
* Women who are 18 years and older.
* There is at least 45 minutes from the time of enrollment to the time patient is transferred to the operating room.

Exclusion Criteria:

* Non-English speaking women.
* Women who are currently pregnant or lactating.
* Women who are hearing impaired.
* Women who have participated in this study before.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Preoperative Anxiety | Day 1: 30 minutes
  The primary variable is anxiety score measured by the State-Trait Anxiety Inventory form Y1 (STAI-Y1) The STAI-Y1 is a 20 item questionnaire which asks subject to rate feelings with a 1-4 pt scale where 1 indicates "not at all" and 4 indicated "very much so". (Range of score 20-80) Higher score equals more anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Thythy Pham, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lee J, Kim HS, Shim KD, Park YS. The Effect of Anxiety, Depression, and Optimism on Postoperative Satisfaction and Clinical Outcomes in Lumbar Spinal Stenosis and Degenerative Spondylolisthesis Patients: Cohort Study. Clin Orthop Surg. 2017 Jun;9(2):177-183. doi: 10.4055/cios.2017.9.2.177. Epub 2017 May 8. PMID 28567219
- [Result] Bradt J, Dileo C, Shim M. Music interventions for preoperative anxiety. Cochrane Database Syst Rev. 2013 Jun 6;2013(6):CD006908. doi: 10.1002/14651858.CD006908.pub2. PMID 23740695
- [Result] Rosen S, Svensson M, Nilsson U. Calm or not calm: the question of anxiety in the perianesthesia patient. J Perianesth Nurs. 2008 Aug;23(4):237-46. doi: 10.1016/j.jopan.2008.05.002. PMID 18657759
- [Result] Wang TF, Wu YT, Tseng CF, Chou C. Associations between dental anxiety and postoperative pain following extraction of horizontally impacted wisdom teeth: A prospective observational study. Medicine (Baltimore). 2017 Nov;96(47):e8665. doi: 10.1097/MD.0000000000008665. PMID 29381942
- [Derived] Chen YB, Barnes H, Westbay L, Wolff B, Shannon M, Adams W, Acevedo-Alvarez M, Mueller ER, Pham TT. Preoperative Music Listening in Pelvic Reconstructive Surgery: A Randomized Trial. Female Pelvic Med Reconstr Surg. 2021 Aug 1;27(8):469-473. doi: 10.1097/SPV.0000000000001070. PMID 34397606